CLINICAL TRIAL: NCT01686516
Title: Methodological Study of Synaptic Plasticity Imaging with Diffusion MRI
Brief Title: Synaptic Plasticity Imaging with Diffusion MRI
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C10-58; 2011-A00034-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2012-09-18 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Brain Aging
Keywords: age; microstructure; diffusion MRI

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diffusion MRI employed in functional imaging has the potential to probe directly brain activation instead of blood changes like the BOLD technique. The researchers investigated these rapid synaptic plasticity changes with visual activation followed by BOLD and diffusion functional MRI as well as anatomical (venography, tractography by diffusion) features in young and aged subjects.

DETAILED DESCRIPTION:
This study is devoted to explore brain plasticity by 2 modes of diffusion weighted imaging (DWI) of the brain :

* functional imaging using DWI and BOLD
* anatomical studies using DWI Theses DWI exams use high b-factor to sample tissue microstructure/metabolism. To correlated these DWI changes with anatomical ones, we used anatomical imaging like T1 maps and susceptibility-based maps.

First, the relatively new technique of diffusion functional magnetic Resonance (DfMRI) was explored to obtain activation of brain following visual stimulations. These modality was compared to BOLD and anatomical venography.

The DWI exams for anatomical (tractography) used both high angular resolution directional diffusion encoding (18 directions) and high b-values (as high as b=12 000 s/mm²) to obtain precise knowledge about tissue microstructure.

Study was approved by the National French Institute of Health and by french organism for biomedical studies (AFFSAPS). Study involve 35 subjects, with 5 additional subjects for eventual rejection because of ineligibility criterion, and compare 15 young (20-30 years) to aged healthy people (60-80 years).

Then, anatomical studies are devoted to obtain microstructures information about brain areas that are changed with age, and to validate fully the feasibility of the DfMRI approach.

ELIGIBILITY:
Inclusion Criteria:

* ages 20-30 years
* 60-80 years

Exclusion Criteria:

* psychological or organic trouble

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: population free of any psychological or organic troubles, with no metal inclusions for MRI convenience.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2012-09-19 (Actual); Study Completion 2012-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm U 825, Toulouse, France, France